CLINICAL TRIAL: NCT05988775
Title: Ipsilateral Transfer of Motor Skill From Lower to Upper Limb in Healthy Adults: a Randomized Controlled Trial
Brief Title: Ipsilateral Transfer of Motor Skill From Lower to Upper Limb in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-HEA-OE-20210610
Record Dates: First submitted 2023-07-30; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-05

CONDITIONS: Healthy
Keywords: ipsilateral transfer; motor performance; lower limb; upper limb; reaching sequence

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Leg training (Experimental): Participants sat on a chair with their left heel resting on the table with the push button switches. participants performed 10 blocks of the aforementioned sequence with their leg, with a 30s break between each block.
  Interventions: Behavioral: Leg training
- Sequence observation (Active Comparator): Participants observed 10 blocks of the sequence with the lights alternating automatically, with a 30s break between each block.
  Interventions: Behavioral: Sequence observation
- Nature movie watching (Other): Participants watched a "scenic relaxation film," for 10 minutes, with a 30s break after every minute.
  Interventions: Other: Nature movie watching

INTERVENTIONS:
Behavioral: Leg training — Participants sat on a chair with their left heel resting on the table with the push button switches. participants performed 10 blocks of the aforementioned sequence with their leg, with a 30s break between each block.
  Arms: Leg training
Behavioral: Sequence observation — Participants observed 10 blocks of the sequence with the lights alternating automatically, with a 30s break between each block.
  Arms: Sequence observation
Other: Nature movie watching — Participants observed 10 blocks of the sequence with the lights alternating automatically, with a 30s break between each block.
  Arms: Nature movie watching

SUMMARY:
To determine whether there is an ipsilateral transfer of motor skill from the lower to the upper limb in healthy adults.

DETAILED DESCRIPTION:
In a single-blind randomized controlled study,45 healthy subjects were randomly allocated to one of three single intervention groups: (1) "Leg Training" group (LT) (15 participants) practiced reaching movement (RM) sequences with the non-dominant left lower limb towards the numbered illuminating switch; (2) "Sequence observation" group (SO) (15 participants) observed the identical sequences of the illuminating switches (Switches Observation (SO) group); and (3) "Nature Movie Watching" (MW) group. (15 participants) watched a neutral nature video. Each subject was asked to attend two consecutive sessions, day after day. The first session included familiarization practice of the motor task, a pretest, a single session intervention (according to group randomization), and a posttest. Subjects participated in two sessions. The second session included a retest, 24 hours after the training. The predefined sequence consisted of six reaching movements in the following order of switches: 1, 4, 3, 5, 4, 2.

Recording apparatus used in tests (pretest, posttest, and retest) and training: A custom-made testing device was set up on a rectangular table with a smooth laminated tabletop of 105 cm × 80 cm and adjustable height. Five switch-led units of 5 cm × 8 cm × 5 cm, each composed of a large push-button switch and a red light-emitting diode (LED), attached to the tabletop in a 38-cm radius half circle, successively numbered from 1 to 5. The system was operated by a desktop computer, interfaced with a data acquisition card of LABVIEW software. The algorithm allowed parameters selection of LED activation (illumination) sequence, duration of RM, the delay between RMs, and the number of RM repetitions. Activation of a specific unit LED was a cue for the subject to reach toward that unit and press the push-button switch. Reaching the switch of an activated unit deactivated it, and the response time, between the activated and deactivated LED, was recorded.

Tests (motor tasks): The non-dominant left arm was tested. Motor task: The subjects performed a sequential movement task on a table with push button switches with lights sequentially turning on to indicate the order. Each switch lit up for 1 second, or until hit. Initially, the participants were required to perform 3 sequences to familiarize themselves with the setup, the task, and the sequence. Then, they performed the pre-test which consisted of two blocks of 5 sequences, i.e. 10 sequences, with a 30s break between blocks. After this, the participants underwent one of the following predetermined interventions groups:

1. "Leg Training" Participants sat on a chair with their left heel resting on the table with the push button switches. They performed 10 blocks of the aforementioned sequence with their leg, with a 30s break between each block.
2. "Sequence observation" Participants observed 10 blocks of the identical sequence with the lights alternating automatically, with a 30s break between each block.
3. "Nature movie watching" Participants watched a "scenic relaxation film" for 10 minutes, with a 30s break after every minute.

Two outcome measures were used: 1. response time (s), 2. failure (%) of the reaching movements, defined as failure to reach the switch in the allotted time (1 sec), or pressing the wrong buzzer.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 35
* right-hand dominant
* healthy according to self-report

Exclusion Criteria:

* musculoskeletal problems or any other problem that may interfere with the performance of the task (extension of an arm or leg while sitting).
* pregnancy

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Change in response time (s) from baseline to post-test | baseline - before the training session, post-test - immediately after the training session
  Average time of movements, measured from the time the switch lights up until it is pressed
Change in response time (s) from post-test to follow up | post-test - immediately after the training session, follow up - 24 hours after the training session
  Average time of movements, measured from the time the switch lights up until it is pressed
Change in response time (s) from baseline to follow up | baseline - before the training session, follow up - 24 hours after the training session
  Average time of movements, measured from the time the switch lights up until it is pressed

SECONDARY OUTCOMES:
Change in failure (%) from baseline to post-test | baseline - before the training session, post-test - immediately after the training session
  Percentage of the reaching movements in which the participant failed to reach the switch in the allotted time (1 sec) or pressed the wrong buzzer.
Change in failure (%) from post-test to follow up | post-test - immediately after the training session, follow up - 24 hours after the training session
  Percentage of the reaching movements in which the participant failed to reach the switch in the allotted time (1 sec) or pressed the wrong buzzer.
Change in failure (%) from base line to follow up | baseline - before the training session, follow up - 24 hours after the training session
  Percentage of the reaching movements in which the participant failed to reach the switch in the allotted time (1 sec) or pressed the wrong buzzer.

CONTACTS AND LOCATIONS:
Overall Officials: Silvi Frenkel-Toledo, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
The datasets (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code generated during and/or analyzed during the current study) will be available from the corresponding author on reasonable request.